CLINICAL TRIAL: NCT05309265
Title: Multidisciplinary Vocational Rehabilitation Intervention to Support the Return to Work of Breast Cancer Patients: a Feasibility Study
Brief Title: Vocational Rehabilitation for the Return to Work of Breast Cancer Patients: a Feasibility Study
Acronym: VocRehab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/0035986
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Cancer Survivors; Return to work; Vocational Rehabilitation; Occupational Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breast cancer patients with work difficulties (Other): Breast cancer patients with work difficulties can receive any of the three types of support, or a combination of these: information, occupational therapy and social support, in order to overcome barriers and return to work/continue to work
  Interventions: Other: Multidisciplinary vocational rehabilitation intervention

INTERVENTIONS:
Other: Multidisciplinary vocational rehabilitation intervention — * Information aims to provide tailored information concerning the work law protection (this support is already provided for all patients, regardless the type of disease, and also for citizens);
  * Occupational therapy aims to facilitate the reintegration in the previous workplace through the development of a rehabilitation intervention to overcome work difficulties in agreement with employee, employer and occupational physician,
  * Social support aims to find new job opportunities (for those who have lost the employment due to the disease) through the giving of support in job search, curriculum preparation, skill analysis, professional retraining and education.

SUMMARY:
In Italy, 50% of new breast cancer (BC) diagnosis occur in female of working age. Although return to work (RTW) is strongly desired by BC patients, cancer survivors are more likely to be unemployed than healthy individuals. Moreover, work difficulties may hindrance this process. Since 2018, the investigators have planned a local social-healthcare pathway which provides a multidisciplinary vocational rehabilitation intervention with the aim to help cancer survivors in their RTW process. To date, the feasibility of the multidisciplinary vocational rehabilitation interventions has not been verified for BC patients.

DETAILED DESCRIPTION:
BC is a public health burden with increasing trends in Western countries. In Italy, 50% of the new BC diagnosis have occurred in female of working age. Even though the return to work (RTW) is strongly desired, cancer survivors are 1.4 times more likely to be unemployed than healthy individuals. Furthermore, work difficulties may occur during this process. To promote the RTW, multidisciplinary interventions have shown moderate quality evidence in cancer survivors.

Since 2018, the investigators have planned a local social-healthcare pathway which provides a multidisciplinary vocational rehabilitation intervention with the aim to help cancer survivors in their RTW process. During the implementation of the pathway, BC patients were referred mainly by the physiotherapists of the Physical Medicine and Rehabilitation Unit (PMRU). As standard care, BC patients can participate to an educational group session held by the physiotherapists after surgery. During this session, work difficulties have emerged.

Thus, the investigators aim to verify the feasibility of the multidisciplinary vocational rehabilitation intervention for a sample of BC patients whit work difficulties who will participate to an educational group session held by the physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer diagnosis (regardless of stage and treatment)
* breast cancer patients in working age
* breast cancer patient who will participate to an educational group session held by the physiotherapists of the PMRU
* breast cancer patients with work difficulties

Exclusion Criteria:

* Breast cancer patients with work issues that cannot be addressed by any of the interventions (e.g., patients who would like to change their job)

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
interception | 12 months
  rate of patients who has been proposed to participate to the feasibility study
acceptation | 12 months
  rate of patients (who has been proposed to participate to the feasibility study) who accept to participate
adherence | 12 months
  rate of patients who participate in the scheduled meeting and in the multidisciplinary intervention proposed; rate of patients who agree to receive the intervention at the workplace (for those eligible)
lost to follow-up | 12 months
  rate of patients who will not attend the scheduled meeting (drop-out rate set ≤ 20%)
satisfaction rate | 12 months
  rate of patients who perceive the modules of the multidisciplinary intervention as supportive for their RTW or work continuation
RTW/work continuation | 12 months
  rate of patients who participate in the study and who will RTW or continued to work

CONTACTS AND LOCATIONS:
Overall Officials: Sara Paltrinieri, Msc OT, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Azienda Unità Sanitaria Locale Reggio Emilia, Reggio Emilia, Reggio Emilia, Italy